CLINICAL TRIAL: NCT04564716
Title: Сlinical Trial of Efficacy, Safety and Immunogenicity of Combined Vector Vaccine Gam-COVID-Vac in SARS-СoV-2 Infection Prophylactic Treatment in Republic of Belarus
Brief Title: Clinical Trial of Efficacy, Safety, and Immunogenicity of Gam-COVID-Vac Vaccine Against COVID-19 in Belarus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Russian Direct Investment Fund (Industry); CRO: iPharma (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 04-Gam-COVID-Vac-2020-RB
Record Dates: First submitted 2020-09-24; First posted 2020-09-25 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: COVID-19; vector vaccine; SARS-CoV-2; adenoviral vector
MeSH Terms: conditions — COVID-19 | interventions — Gam-COVID-Vac vaccine

STUDY DESIGN:
Intervention Model Description: Randomized double-blind placebo-controlled
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Group (Experimental): Gam-COVID-Vac combined vector vaccine, 0,5ml/dose+0,5 ml/dose prime-boost immunization in days 1 (component I rAd26-S) and 21(component II rAd5-S)
  Interventions: Biological: Gam-COVID-Vac
- Control Group (Placebo Comparator): placebo, 0,5ml/dose+0,5 ml/dose immunization in days 1 and 21
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Gam-COVID-Vac — vaccine for intramuscular injection
  Arms: Primary Group
Other: Placebo — placebo comparator
  Arms: Control Group

SUMMARY:
Randomized, double-blind (blinded for the trial subject and the study physician), placebo controlled, multi-center clinical trial in parallel assignment of efficacy, immunogenicity, and safety of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection in adults in the SARS-СoV-2 infection prophylactic treatment.

DETAILED DESCRIPTION:
Overall of 110 volunteers aged 18 to 60 should be screened taking into account possible early departure from the study. It is supposed that 100 subjects will complete all screening procedures and will be randomized in a 3:1 ratio into two groups: a control group (using placebo, 25 subjects) and a study group (using Gam-COVID-Vac Combined Vector Vaccine to Prevent Coronavirus Infection Caused by SARS-CoV-2", 75 subjects).

The duration of participation in the study for one subject will be 180±14 days after the first dose of IMP/placebo, during which each subject will undergo a screening visit and five face-to-face visits to the doctor-researcher. Intramuscular injection of IMP or placebo will be carried out on vaccination visits N 1 and N 2 (Day 0 and Day 21±2). Further observation visits No 3, 4, 5 will be conducted on days 28±2, 42±2 and 180±14 respectively. It is allowed to conduct observation visits No. 3, 4 via telephone contact (TC). During the monitoring visits, all subjects of the study will be assessed on key vital indicators and data will be collected on changes in the status and well-being of the subjects since the previous visit.

The duration of participation in the study for one subject will be 180±14 days after the first dose of IMP/placebo, during which each subject will undergo a screening visit and five observation visits. Intramuscular injection of IMP or placebo will be carried out on vaccination visits N 1 and N 2 (Day 0 and Day 21±2). Further observation visits No 3, 4, 5 will be conducted on days 28±2, 42±2 and 180±14 respectively.

ELIGIBILITY:
Inclusion Criteria:

* The subject's written informed consent to participate in the study;
* Male and female subjects between the ages of 18 and 60 years (inclusive).
* A negative test result for HIV, hepatitis, syphilis;
* Negative result of research on antibodies IgM and IgG to SARS Cov2 by enzyme-linked immunosorbent assay;
* A negative result of the COVID-2019 study, as determined by the PCR method at the screening visit;
* Lack of COVID-2019 in anamnesis;
* Lack of contact of the subject with COVID-2019 patients for at least 14 days before inclusion in the study (according to the participant);
* Agreement to use effective contraceptive methods throughout the study period;
* Negative pregnancy test based on the results of a urine test at a screening visit (for women of childbearing age);
* A negative test for the presence of narcotic substances and psycho-stimulating drugs in the urine at the screening visit;
* Negative alcohol test at the screening visit;
* Lack of pre-existing post-vaccination reactions or post-vaccination complications following the use of immunobiological drugs;
* No acute infectious and/or respiratory diseases for at least 14 days before inclusion in the study.

Exclusion Criteria:

* Any vaccination/immunization carried out within 30 days prior to enrollment in the study;
* Treatment with steroids (except hormonal contraceptives) and/or with immunoglobulins or other blood products not completed 30 days before inclusion in the study;
* Immunosuppressive therapy completed less than three months before inclusion in the study;
* Female subjects during pregnancy or breastfeeding;
* Acute coronary syndrome or stroke suffered less than one year before inclusion into the study;
* Tuberculosis, chronic systemic infections;
* Aggravated allergy anamnesis (anamnesis of anaphylactic shock, Quinque edema, polymorphic exudative eczema, atopia, serum disease), hypersensitivity or allergic reactions to immunobiological drugs, known allergic reactions to the components of the drug, aggravation of allergic diseases on the day of inclusion in the study;
* The presence of neoplasms in the anamnesis (codes C00-D09);
* Donated blood or plasma (450 ml or more) less than 2 months before inclusion in the study;
* Splenectomy in anamnesis;
* Neutropenia (decrease in absolute number of neutrophils less than 1000/mm3), agraneulocytosis, significant haemorrhage, severe anaemia (hemoglobin less than 80 g/l), immunodeficiency in anamnesis for 6 months before inclusion in the study;
* Subjects with an active form of disease caused by human immunodeficiency virus, syphilis, hepatitis B and C;
* Anorexia, protein deficiency of any origin;
* Chronic autoimmune diseases or systemic collagenoses in anamnesis
* Extensive tattoos at the injection site (deltoid region) that do not allow for an assessment of the local response to IMP/placebo administration;
* Alcoholism and drug addiction in anamnesis;
* Participation of the subject in any other interventional clinical trial;
* Any other condition of the subject which, in the opinion of the researcher's medical practitioner, may prevent completion of the investigation according to the protocol;
* Staff of research centers and other staff directly involved in the study and their families.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-03-28 (Estimated); Study Completion 2021-04-10 (Estimated)

PRIMARY OUTCOMES:
percentage of trial subjects with coronavirus disease 2019 (COVID-19) developed within 6 months after the first dose | through the whole study, an average of 180 days
  Demonstrate the superiority of Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection compared to placebo, based on the percentage of trial subjects with coronavirus disease 2019 (COVID-19) developed within 6 months after the second dose of the study drug/placebo, as confirmed with the method of polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
the severity of the clinical course of COVID-19 | through the whole study, an average of 180 days
  Assess the efficacy of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus compared to placebo, based on the severity of the clinical course of COVID-19
Changing of antibody levels against the SARS-CoV-2 glycoprotein S | day before injecting the first dose of the study drug/placebo and 42±2 and 180±14 days after the first dose
  Assess the immunogenicity of the Gam-COVID-Vac combined vector vaccine against the SARS-CoV-2-induced coronavirus infection compared to placebo, based on the geometric mean titer of SARS-CoV-2 glycoprotein-specific antibodies
Incidence of adverse events in trial subjects | through the whole study, an average of 180 days
  Incidence of adverse events in trial subjects compared to placebo
Severity of adverse events in trial subjects | through the whole study, an average of 180 days
  Severity of adverse events in trial subjects compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Roman Plotnikov, Study Chair — CRO: iPharma
Locations (8):
- Belarus (8):
  - Health Institution "14th Central Regional Polyclinic of the Partisan district of Minsk", Minsk
  - Health Institution "19th Central Regional Polyclinic of the Pervomaysk district of Minsk", Minsk
  - Health Institution "1st Central Regional Clinical Polyclinic of the Central district of Minsk", Minsk
  - Health Institution "28th Regional Polyclinic of Minsk", Minsk
  - Health Institution "4th City Polyclinic of Minsk", Minsk
  - Health Institution "5th City Clinical Polyclinic of Minsk", Minsk
  - Health Institution "Minsk Order of the Red Banner of Labor Regional Clinical Hospital, Minsk
  - Health Institution "Vitebsk Regional Clinical Hospital", Vitebsk